CLINICAL TRIAL: NCT02808429
Title: A Phase II Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Atacicept in IgA Nephropathy
Brief Title: Efficacy and Safety of Atacicept in IgA Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early as per sponsor decision due to unexpectedly slow enrollment.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS700461-0035; 2016-002262-31 (EudraCT Number)
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-01

CONDITIONS: IgA Nephropathy
Keywords: Atacicept; IgA Nephropathy; Berger´s disease; Glomerulonephritis; Proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis; Proteinuria | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental)
  Interventions: Drug: Placebo
- Atacicept 25 mg (Experimental)
  Interventions: Drug: Atacicept 25 mg
- Atacicept 75 mg (Experimental)
  Interventions: Drug: Atacicept 75 mg

INTERVENTIONS:
Drug: Placebo — Participants received placebo matched to Atacicept once weekly as subcutaneous (SC) injection during this study up to a maximum of 72.1 weeks.
  Arms: Placebo
Drug: Atacicept 25 mg — Participants received 25 milligrams (mg) of Atacicept once weekly as SC injection during this study up to a maximum of 73.6 weeks.
  Arms: Atacicept 25 mg
Drug: Atacicept 75 mg — Participants received 75 mg of Atacicept once weekly as SC injection during this study up to a maximum of 74.1 weeks.
  Arms: Atacicept 75 mg

SUMMARY:
This main purpose of this study was to evaluate the safety, tolerability, dose response and efficacy of Atacicept in participants with IgA nephropathy and persistent proteinuria. The study hypothesis was that treatment with Atacicept would reduce proteinuria compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to (>=)18 years of age
* Biopsy-proven Immunoglobulin (IgA) nephropathy
* Urine Protein to Creatinine Ratio (UPCR) >= 0.75 and <= 6 milligram per milligram (mg/mg) during screening
* Stable and optimal dose of Angiotensin converting enzyme (ACE) inhibitor and/or angiotensin II receptor blockers (ARB) at least 8 weeks prior to screening

Exclusion Criteria:

* Concomitant significant renal disease other than IgA nephropathy
* IgA nephropathy with significant glomerulosclerosis or cortical scarring
* Diagnosis of Henoch-Schonlein purpura
* Failure to meet estimated glomerular filtration rate (eGFR) and biopsy requirement criteria
* Serum IgG below 6 grams per liter (g/L)
* Use of cyclophosphamide ever or use of other immunosuppressants or systemic corticosteroids within 4 months
* Active infection requiring hospitalization or treatment with parenteral anti-infectives within 4 weeks
* History, or current diagnosis, of active tuberculosis (TB), or untreated latent TB infection
* History of or positive HIV and/or positive for hepatitis B or Hepatitis C at screening
* History of malignancy
* Nursing or pregnancy
* Any condition, including any uncontrolled disease state other than IgA nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (18):
- United States (16):
  - AKDHC Medical Research Services, LLC., Glendale, Arizona
  - California Institute of Renal Research - Chula Vista Location, Chula Vista, California
  - Colorado Kidney Care PC - Dr. Marder, Denver, Colorado
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - GA Nephrology Associates, Lawrenceville, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Ohio State University Clinical Trials Management Office - Ohio State CTMO Parent, Columbus, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Nephrotex Research Group, Dallas, Texas
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
- Juntendo University Hospital - Dept of Nephrology/Hypertension, Bunkyō City, Japan
- University Hospitals of Leicester NHS Trust - ULTIMATE PARENT, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website.
URL: https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: US Medical Information website, Medical Resources — http://medical.emdserono.com/en_US/home.html
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700461-0035

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was to be conducted in 2 parts; Part A and Part B. However, study was terminated early as per sponsor decision due to unexpectedly slow enrollment and Part B was not initiated.
Period: Overall Study
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Started | 5 | 6 | 5
Completed | 2 | 5 | 3
Not Completed | 3 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Premature study termination by sponsor | 2 | 0 | 1
Not completed — Relocation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all randomized participants who had received at least 1 dose of the Investigational Medicinal Product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Total
Number analyzed (Participants) | 5 | 6 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (3.1) | 41 (16.9) | 43 (8.7) | 43 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 2 | 8
  Male | 4 | 1 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 4
  Not Hispanic or Latino | 5 | 5 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 5 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs), Adverse Event of Special Interest (AESIs), Serious TEAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: Adverse Event (AE): any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE: AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: AEs that developed or worsened/became serious during on-treatment period (time from the first dose of study drug up to the end of study [Week 96]). TEAEs included serious AEs and non- serous AEs. AESIs included infections, cardiac failure, cardiomyopathy/ ischemic heart disease, hypersensitivity reaction (including anaphylactic/anaphylactoid shock conditions, asthma/bronchospasm, and angioedema), injection site reactions (ISRs) and demyelinating disorders. Investigator or his /her designee assessed ISRs as local reactions (redness, bruising, swelling, induration and itching).
Time Frame: Baseline up to 96 weeks
Population: The safety population set (SAF) included all randomized participants who received at least 1 dose of IMP and had at least one post-dose assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
percentage of participants
  Participants with TEAE | 100 | 100 | 60
  Participants with AESI: Cardiac failure | 0 | 0 | 0
  Participants with AESI: Ischaemic heart disease | 0 | 0 | 0
  Participants with AESI: Cardiac arrhythmia | 0 | 0 | 0
  Partcipants with AESI: Hypersensitivity reactions | 20 | 66.67 | 20
  Partcipants with AESI: Demyalinating disorders | 0 | 0 | 0
  Partcipants with AESI: Injection site reactions | 0 | 83.3 | 60
  Partcipants with AESI: Infections | 40 | 83.33 | 20
  Participants with serious TEAEs | 20 | 50 | 0
  Participants with TEAEs leading to discontinuation | 0 | 16.66 | 0
  Participants with TEAEs leading to death | 0 | 0 | 0

2. Secondary Outcome: Serum Atacicept Concentrations
Description: Serum Atacicept Concentrations was to be performed; however; as per changed in planned analysis the outcome measure related to pharmacokinetic parameters was not assessed.
Time Frame: Week 0 Day 1 (pre-dose), Weeks 1, 2, 4, 8, 12, 16, 24, 40, 48, 72, Early Termination (up to Week 72) and Post-treatment (PT) Follow Up (FU) Weeks 4, 12 and 24
Population: As per changed in planned analysis the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline Levels in Serum Immunoglobulin A (IgA)
Description: The change in serum levels of IgA from baseline was reported.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, Early Termination (up to Week 72) and PT FU Weeks 4, 12 and 24
Population: The safety population set (SAF) included all randomized participants who received at least 1 dose of IMP and had at least one post-dose assessment. Here "number analyzed" = participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
gram per liter
  Change at Week 1 | -0.194 (0.3012) | -0.203 (0.1325) | -0.278 (0.1561)
  Change at Week 2 | -0.114 (0.2825) | -0.280 (0.1108) | -0.486 (0.2289)
  Change at Week 4 | -0.014 (0.3570) | -0.197 (0.1952) | -0.828 (0.2319)
  Change at Week 8: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 8 | 0.008 (0.5340) | -0.572 (0.2838) | -1.144 (0.4997)
  Change at Week 12: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 12 | -0.030 (0.4011) | -0.476 (0.3879) | -1.146 (0.4226)
  Change at Week 16: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 16 | 0.044 (0.4869) | -0.692 (0.3608) | -1.296 (0.4237)
  Change at Week 20: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 20 | 0.218 (0.6157) | -0.616 (0.2880) | -1.430 (0.4635)
  Change at Week 24: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 24 | 0.212 (0.3140) | -0.514 (0.4552) | -1.424 (0.5226)
  Change at Week 32: number analyzed (Participants) | 5 | 4 | 5
  Change at Week 32 | 0.180 (0.4924) | -0.920 (0.2950) | -1.468 (0.3851)
  Change at Week 40: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 40 | 0.112 (0.7745) | -0.963 (0.2815) | -1.388 (0.3212)
  Change at Week 48: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 48 | 0.526 (1.2935) | -0.710 (0.3804) | -1.375 (0.4680)
  Change at Week 60: number analyzed (Participants) | 4 | 3 | 4
  Change at Week 60 | 0.233 (0.3676) | -0.733 (0.3057) | -1.283 (0.4308)
  Change at Week 72: number analyzed (Participants) | 3 | 3 | 3
  Change at Week 72 | 0.307 (0.3650) | -0.957 (0.2157) | -1.240 (0.4491)
  Change at Early termination: number analyzed (Participants) | 2 | 3 | 2
  Change at Early termination | 0.420 (0.0849) | -0.493 (0.2173) | -1.835 (0.1344)
  Change at PT FU Week 4: number analyzed (Participants) | 5 | 5 | 3
  Change at PT FU Week 4 | 0.300 (0.4757) | -0.452 (0.3529) | -1.223 (0.2515)
  Change at PT FU Week 12: number analyzed (Participants) | 5 | 5 | 4
  Change at PT FU Week 12 | 0.622 (0.7436) | -0.440 (0.6335) | -0.668 (0.2843)
  Change at PT FU Week 24: number analyzed (Participants) | 4 | 5 | 4
  Change at PT FU Week 24 | 0.563 (0.6716) | -0.420 (0.6503) | -0.370 (0.1160)

4. Secondary Outcome: Change From Baseline Levels in Serum Iimmunoglobulin G (IgG)
Description: The change in serum levels of IgG from baseline was reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
gram per liter
  Change at Week 1 | -0.630 (0.5524) | -0.480 (0.4289) | -0.444 (0.4372)
  Change at Week 2 | -0.362 (0.7146) | -0.650 (0.5764) | -0.898 (0.5507)
  Change at Week 4 | -0.354 (0.7073) | -0.415 (0.4965) | -1.792 (0.8182)
  Change at Week 8: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 8 | -0.562 (1.0023) | -1.128 (0.3574) | -2.812 (1.2085)
  Change at Week 12: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 12 | -0.472 (0.9304) | -0.930 (0.7748) | -3.126 (0.9324)
  Change at Week 16: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 16 | -0.608 (1.1858) | -1.480 (0.4687) | -3.360 (0.8546)
  Change at Week 20: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 20 | 0.016 (1.0781) | -1.024 (0.3893) | -3.684 (0.7597)
  Change at Week 24: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 24 | -0.748 (1.0059) | -0.926 (0.8289) | -3.776 (1.0876)
  Change at Week 32: number analyzed (Participants) | 5 | 4 | 5
  Change at Week 32 | -0.296 (1.1195) | -1.055 (0.5701) | -3.962 (0.8830)
  Change at Week 40: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 40 | 0.218 (0.8904) | -1.363 (0.4895) | -3.623 (0.2993)
  Change at Week 48: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 48 | 0.256 (1.5731) | -0.600 (0.7654) | -3.745 (0.4608)
  Change at Week 60: number analyzed (Participants) | 4 | 3 | 4
  Change at Week 60 | 0.305 (1.2881) | -0.743 (1.5627) | -3.368 (0.5721)
  Change at Week 72: number analyzed (Participants) | 3 | 3 | 3
  Change at Week 72 | -0.203 (1.3606) | -0.867 (0.7772) | -3.477 (0.8618)
  Change at Early Termination: number analyzed (Participants) | 2 | 3 | 2
  Change at Early Termination | 0.655 (0.5445) | -1.547 (0.5353) | -3.995 (0.0636)
  Change at PT FU Week 4: number analyzed (Participants) | 5 | 5 | 3
  Change at PT FU Week 4 | 0.360 (1.7711) | -0.736 (0.7900) | -2.553 (0.7160)
  Change at PT FU Week 12: number analyzed (Participants) | 5 | 5 | 4
  Change at PT FU Week 12 | 0.922 (1.2793) | -0.800 (1.4692) | -1.300 (0.5610)
  Change at PT FU Week 24: number analyzed (Participants) | 4 | 5 | 4
  Change at PT FU Week 24 | 0.273 (0.9758) | -0.878 (1.0395) | 0.020 (1.2498)

5. Secondary Outcome: Change From Baseline Levels in Serum Immunoglobulin M (IgM)
Description: The change in serum levels of IgM from baseline was reported.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, Early Termination (up to Week 72) and at PT FU Weeks 4, 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
gram per liter
  Change at Week 1 | -0.082 (0.0835) | -0.072 (0.0736) | -0.096 (0.0924)
  Change at Week 2 | -0.054 (0.1026) | -0.140 (0.1906) | -0.102 (0.1625)
  Change at Week 4 | -0.002 (0.1190) | -0.197 (0.2655) | -0.410 (0.1637)
  Change at Week 8: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 8 | 0.006 (0.1710) | -0.302 (0.3114) | -0.558 (0.1859)
  Change at Week 12: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 12 | 0.022 (0.0955) | -0.360 (0.3169) | -0.638 (0.2497)
  Change at Week 16: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 16 | 0.024 (0.1412) | -0.408 (0.3531) | -0.710 (0.2463)
  Change at Week 20: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 20 | 0.082 (0.2288) | -0.444 (0.3965) | -0.748 (0.2500)
  Change at Week 24: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 24 | -0.016 (0.1390) | -0.364 (0.3377) | -0.774 (0.2517)
  Change at Week 32: number analyzed (Participants) | 5 | 4 | 5
  Change at Week 32 | -0.016 (0.1566) | -0.510 (0.4498) | -0.796 (0.2773)
  Change at Week 40: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 40 | 0.036 (0.1464) | -0.247 (0.1553) | -0.848 (0.2668)
  Change at Week 48: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 48 | 0.012 (0.1951) | -0.227 (0.1250) | -0.848 (0.2557)
  Change at Week 60: number analyzed (Participants) | 4 | 3 | 4
  Change at Week 60 | -0.033 (0.0907) | -0.297 (0.2495) | -0.843 (0.2573)
  Change at Week 72: number analyzed (Participants) | 3 | 3 | 3
  Change at Week 72 | -0.027 (0.0153) | -0.337 (0.2914) | -0.900 (0.3081)
  Change at Early Termination: number analyzed (Participants) | 2 | 3 | 2
  Change at Early Termination | 0.115 (0.0354) | -0.463 (0.1626) | -0.670 (0.1414)
  Change at PT FU Week 4: number analyzed (Participants) | 5 | 5 | 3
  Change at PT FU Week 4 | -0.048 (0.1941) | -0.328 (0.1906) | -0.667 (0.2259)
  Change at PT FU Week 12: number analyzed (Participants) | 5 | 5 | 4
  Change at PT FU Week 12 | 0.058 (0.2281) | -0.214 (0.1739) | -0.465 (0.2319)
  Change at PT FU Week 24: number analyzed (Participants) | 4 | 5 | 4
  Change at PT FU Week 24 | 0.020 (0.1687) | -0.178 (0.1504) | -0.340 (0.1896)

6. Secondary Outcome: Change From Baseline in Serum Galactose Deficient-IgA1 (Gd-IgA1) Levels
Description: The change in serum Gd-IgA1 from baseline was reported.
Time Frame: Baseline, Weeks 4, 12, 24, 48, 72, Early Termination (up to Week 72 and at PT FU Weeks 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
nanogram per milliliter (ng/mL)
  Change at Week 4 | -1438 (598.2) | -620 (1580.4) | -2288 (730.5)
  Change at Week 12: number analyzed (Participants) | 5 | 5 | 5
  Change at Week 12 | -380 (1505.0) | -1672 (1459.2) | -2778 (1345.8)
  Change at Week 24: number analyzed (Participants) | 5 | 5 | 4
  Change at Week 24 | 160 (848.8) | -1912 (1835.0) | -3660 (1940.9)
  Change at Week 48: number analyzed (Participants) | 5 | 3 | 4
  Change at Week 48 | 1140 (4339.5) | -423 (795.1) | -2938 (1756.9)
  Change at Week 72: number analyzed (Participants) | 3 | 3 | 3
  Change at Week 72 | 580 (2594.8) | -1327 (1181.4) | -3202 (1594.9)
  Change at Early Termination: number analyzed (Participants) | 2 | 3 | 2
  Change at Early Termination | 3520 (4638.6) | -2383 (2551.1) | -2680 (1258.7)
  Change at PT FU Week 12: number analyzed (Participants) | 5 | 5 | 3
  Change at PT FU Week 12 | 1926 (3523.3) | -772 (2050.2) | -818 (1277.9)
  Change at PT FU Week 24: number analyzed (Participants) | 3 | 5 | 2
  Change at PT FU Week 24 | 1673 (5072.9) | -1262 (2444.1) | -1090 (70.7)

7. Secondary Outcome: Change From Baseline in Serum Complement C3 and C4 Levels
Description: The change in serum component C3 and C4 from baseline were reported.
Time Frame: Baseline, Week 12, 24, 48, 72, Early Termination (up to Week 72) and at PT FU Weeks 12 and 24
Population: The safety population set (SAF) consisted of all randomized participants who received at least 1 dose of IMP and had at least one post-dose assessment. "Number of participants analyzed" signifies participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: milligram per liter
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 5 | 5
milligram per liter
  Complement C3: Change at Week 12 | -60.0 (88.32) | 80.0 (125.10) | 122.0 (114.76)
  Complement C3: Change at Week 24: number analyzed (Participants) | 5 | 5 | 4
  Complement C3: Change at Week 24 | -38.0 (100.85) | -6.0 (220.64) | 70.0 (104.24)
  Complement C3: Change at Week 48: number analyzed (Participants) | 5 | 3 | 4
  Complement C3: Change at Week 48 | 82.0 (215.57) | 63.3 (110.15) | 162.5 (219.91)
  Complement C3: Change at Week 72: number analyzed (Participants) | 3 | 3 | 3
  Complement C3: Change at Week 72 | -56.7 (127.41) | 43.3 (212.21) | 196.7 (196.55)
  Complement C3: Change at Early Termination: number analyzed (Participants) | 2 | 3 | 1
  Complement C3: Change at Early Termination | -145.0 (190.92) | -60.0 (284.78) | 180.0
  Complement C3: Change at PT FU Week 12: number analyzed (Participants) | 5 | 5 | 3
  Complement C3: Change at PT FU Week 12 | -12.0 (106.16) | -96.0 (196.67) | 170.0 (390.00)
  Complement C3: Change at PT FU Week 24: number analyzed (Participants) | 4 | 5 | 4
  Complement C3: Change at PT FU Week 24 | -85.0 (183.76) | -144.0 (93.97) | 164.0 (205.45)
  Complement C4: Change at Week 12 | -26.8 (25.35) | 13.4 (9.24) | 33.8 (44.81)
  Complement C4: Change at Week 24: number analyzed (Participants) | 5 | 5 | 4
  Complement C4: Change at Week 24 | -27.0 (32.26) | 8.8 (29.66) | 34.3 (40.20)
  Complement C4: Change at Week 48: number analyzed (Participants) | 5 | 3 | 4
  Complement C4: Change at Week 48 | -0.4 (20.74) | 33.3 (18.90) | 16.0 (27.89)
  Complement C4: Change at Week 72: number analyzed (Participants) | 3 | 3 | 3
  Complement C4: Change at Week 72 | -43.0 (82.46) | 12.0 (17.35) | 49.7 (30.02)
  Complement C4: Change at Early Termination: number analyzed (Participants) | 2 | 3 | 1
  Complement C4: Change at Early Termination | -22.0 (32.53) | -8.0 (38.57) | 125.0
  Complement C4: Change at PT FU Week 12: number analyzed (Participants) | 5 | 5 | 3
  Complement C4: Change at PT FU Week 12 | -12.6 (32.00) | -4.2 (9.07) | -1.3 (44.52)
  Complement C4: Change at PT FU Week 24: number analyzed (Participants) | 4 | 5 | 4
  Complement C4: Change at PT FU Week 24 | -37.0 (64.97) | -18.2 (30.34) | 19.5 (18.30)

8. Secondary Outcome: Change From Baseline in Immune Cell Subsets by Flow Cytometry Analysis
Description: Change from baseline in immune cell subsets included total T cells, helper T cells, cytotoxic T cells, total B cells (assay with [AW] CD45 or assay without [AWO] CD45), mature naïve B cells, memory B cells, plasma cells, plasma blasts, and natural killer (NK) cells and were reported. Analysis was performed by flow cytometry analysis.
Time Frame: Baseline, Weeks 4, 12, 24, 48, 72, Early Termination (up to Week 72) and at PT FU Week 24
Population: Flow Cytometry (FC) Set: all participants in SAF set who were part of the selected sites for FC analysis and who had at least 1 sample taken for FC analysis. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure. and "number analyzed" signifies those participants who were evaluable for specified category.
Measure: Mean (Standard Deviation); unit: cells per microliter
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 2 | 2 | 3
cells per microliter
  Cytotoxic T Cells: Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  Cytotoxic T Cells: Change at Week 4 |  | -22.5 (215.67) | 46.7 (72.57)
  Cytotoxic T Cells: Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  Cytotoxic T Cells: Change at Week 12 | 713.0 | -114.0 | 75.0 (33.41)
  Cytotoxic T Cells: Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  Cytotoxic T Cells: Change at Week 24 | 101.5 (243.95) | -30.5 (125.16) | 37.0 (39.60)
  Cytotoxic T Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Cytotoxic T Cells: Change at Week 48 | 9.0 (224.86) |  | 38.0 (42.43)
  Cytotoxic T Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 2
  Cytotoxic T Cells: Change at Week 72 | -60.0 |  | -186.0 (289.91)
  Cytotoxic T Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 1
  Cytotoxic T Cells: Change at Early Termination | 282.0 |  | 45.0
  Cytotoxic T Cells: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Cytotoxic T Cells: Change at PT FU Week 24 | 132.0 |  |
  Helper T Cells: Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  Helper T Cells: Change at Week 4 |  | 59.0 (240.42) | 114.7 (117.05)
  Helper T Cells: Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  Helper T Cells: Change at Week 12 | 124.0 | -51.0 | 221.3 (85.33)
  Helper T Cells: Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  Helper T Cells: Change at Week 24 | -79.0 (190.92) | 134.0 (124.45) | 85.0 (45.25)
  Helper T Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Helper T Cells: Change at Week 48 | -129.5 (338.70) |  | 72.5 (86.97)
  Helper T Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 2
  Helper T Cells: Change at Week 72 | -170.0 |  | -312.5 (427.80)
  Helper T Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 1
  Helper T Cells: Change at Early Termination | 81.0 |  | 348.0
  Helper T Cells: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Helper T Cells: Change at PT FU Week 24 | 90.0 |  |
  Mature naive B Cells: Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  Mature naive B Cells: Change at Week 4 |  | -76.5 (12.02) | -17.0 (78.31)
  Mature naive B Cells: Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  Mature naive B Cells: Change at Week 12 | 137.0 | -106.0 | -14.7 (94.07)
  Mature naive B Cells: Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  Mature naive B Cells: Change at Week 24 | 1.0 (42.43) | -117.5 (51.62) | -87.5 (109.60)
  Mature naive B Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Mature naive B Cells: Change at Week 48 | 21.5 (74.25) |  | -91.0 (107.48)
  Mature naive B Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  Mature naive B Cells: Change at Week 72 | -24.0 |  | -32.0
  Mature naive B Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 1
  Mature naive B Cells: Change at Early Termination | 36.0 |  | -1.0
  Mature naive B Cells: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Mature naive B Cells: Change at PT FU Week 24 | 8.0 |  |
  Memory B Cells: Change at Week 4: number analyzed (Participants) | 0 | 1 | 2
  Memory B Cells: Change at Week 4 |  | 8.0 | 14.5 (2.12)
  Memory B Cells: Change at Week 12: number analyzed (Participants) | 1 | 0 | 2
  Memory B Cells: Change at Week 12 | 5.0 |  | 34.0 (0.00)
  Memory B Cells: Change at Week 24: number analyzed (Participants) | 2 | 1 | 2
  Memory B Cells: Change at Week 24 | -1.5 (7.78) | 13.0 | 5.5 (21.92)
  Memory B Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Memory B Cells: Change at Week 48 | -1.0 (4.24) |  | 5.0 (16.97)
  Memory B Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  Memory B Cells: Change at Week 72 | -6.0 |  | 8.0
  Memory B Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 0
  Memory B Cells: Change at Early Termination | -3.0 |  |
  Memory B Cells: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Memory B Cells: Change at PT FU Week 24 | 6.0 |  |
  NK Cells: Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  NK Cells: Change at Week 4 |  | 19.0 (227.69) | 88.3 (30.62)
  NK Cells: Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  NK Cells: Change at Week 12 | 43.0 | -105.0 | 74.0 (89.94)
  NK Cells: Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  NK Cells: Change at Week 24 | 44.5 (20.51) | -34.5 (112.43) | 37.5 (58.69)
  NK Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  NK Cells: Change at Week 48 | 20.5 (16.26) |  | 39.0 (48.08)
  NK Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  NK Cells: Change at Week 72 | 130.0 |  | 104.0
  NK Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 1
  NK Cells: Change at Early Termination | 54.0 |  | 12.0
  NK Cells:Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  NK Cells:Change at PT FU Week 24 | 81.0 |  |
  Plasma Blasts: Change at Week 4: number analyzed (Participants) | 0 | 1 | 2
  Plasma Blasts: Change at Week 4 |  | 0.10 | -0.05 (0.071)
  Plasma Blasts: Change at Week 12: number analyzed (Participants) | 1 | 0 | 2
  Plasma Blasts: Change at Week 12 | -0.10 |  | 0.55 (0.212)
  Plasma Blasts: Change at Week 24: number analyzed (Participants) | 2 | 1 | 2
  Plasma Blasts: Change at Week 24 | 0.05 (0.071) | -0.30 | 0.10 (0.283)
  Plasma Blasts: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Plasma Blasts: Change at Week 48 | 1.40 (1.414) |  | 0.15 (0.212)
  Plasma Blasts: Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  Plasma Blasts: Change at Week 72 | -0.10 |  | 0.40
  Plasma Blasts: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 0
  Plasma Blasts: Change at Early Termination | 0.80 |  |
  Plasma Blasts: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Plasma Blasts: Change at PT FU Week 24 | 3.40 |  |
  Plasma Cells: Change at Week 4: number analyzed (Participants) | 0 | 1 | 2
  Plasma Cells: Change at Week 4 |  | 0.10 | 0.00 (0.141)
  Plasma Cells: Change at Week 12: number analyzed (Participants) | 1 | 0 | 2
  Plasma Cells: Change at Week 12 | -0.10 |  | 0.15 (0.212)
  Plasma Cells: Change at Week 24: number analyzed (Participants) | 2 | 1 | 2
  Plasma Cells: Change at Week 24 | 0.05 (0.071) | -0.10 | 0.00 (0.000)
  Plasma Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Plasma Cells: Change at Week 48 | 0.30 (0.283) |  | 0.00 (0.000)
  Plasma Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  Plasma Cells: Change at Week 72 | 0.00 |  | 0.20
  Plasma Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 0
  Plasma Cells: Change at Early Termination | 0.20 |  |
  Plasma Cells: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Plasma Cells: Change at PT FU Week 24 | 0.10 |  |
  Total B cells (AW CD45): Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  Total B cells (AW CD45): Change at Week 4 |  | -50.0 (36.77) | 37.3 (64.39)
  Total B cells (AW CD45): Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  Total B cells (AW CD45): Change at Week 12 | 154.0 | -105.0 | 108.7 (88.90)
  Total B cells (AW CD45): Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  Total B cells (AW CD45): Change at Week 24 | -0.5 (57.28) | -78.0 (131.52) | -32.5 (116.67)
  Total B cells (AWh CD45): Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Total B cells (AWh CD45): Change at Week 48 | 20.0 (91.92) |  | -27.5 (115.26)
  Total B cells (AW CD45): Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  Total B cells (AW CD45): Change at Week 72 | -31.0 |  | 2.0
  Total B cells (AW CD45): Change at Early Termination: number analyzed (Participants) | 1 | 0 | 1
  Total B cells (AW CD45): Change at Early Termination | 43.0 |  | 71.0
  Total B cells (AW CD45): Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Total B cells (AW CD45): Change at PT FU Week 24 | 27.0 |  |
  Total B cells (AWO CD45): Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  Total B cells (AWO CD45): Change at Week 4 |  | -33.0 (104.65) | 41.0 (40.60)
  Total B cells (AWO CD45): Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  Total B cells (AWO CD45): Change at Week 12 | 16.0 | -137.0 | 52.0 (65.09)
  Total B cells (AWO CD45): Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  Total B cells (AWO CD45): Change at Week 24 | -11.0 (53.74) | -96.5 (135.06) | -40.5 (88.39)
  Total B cells (AWO CD45): Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Total B cells (AWO CD45): Change at Week 48 | 9.0 (113.14) |  | -52.5 (81.32)
  Total B cells (AWO CD45): Change at Week 72: number analyzed (Participants) | 1 | 0 | 1
  Total B cells (AWO CD45): Change at Week 72 | -38.0 |  | -78.0
  Total B cells (AWO CD45): Change at Week Early Termination: number analyzed (Participants) | 1 | 0 | 1
  Total B cells (AWO CD45): Change at Week Early Termination | 23.0 |  | 48.0
  Total B cells (AWO CD45): Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Total B cells (AWO CD45): Change at PT FU Week 24 | -36.0 |  |
  Total T Cells: Change at Week 4: number analyzed (Participants) | 0 | 2 | 3
  Total T Cells: Change at Week 4 |  | 40.0 (466.69) | 169.0 (189.71)
  Total T Cells: Change at Week 12: number analyzed (Participants) | 1 | 1 | 3
  Total T Cells: Change at Week 12 | 861.0 | -165.0 | 314.7 (50.54)
  Total T Cells: Change at Week 24: number analyzed (Participants) | 2 | 2 | 2
  Total T Cells: Change at Week 24 | 18.5 (419.31) | 111.0 (260.22) | 130.0 (2.83)
  Total T Cells: Change at Week 48: number analyzed (Participants) | 2 | 0 | 2
  Total T Cells: Change at Week 48 | -116.5 (564.98) |  | 113.5 (140.71)
  Total T Cells: Change at Week 72: number analyzed (Participants) | 1 | 0 | 2
  Total T Cells: Change at Week 72 | -227.0 |  | -529.5 (767.21)
  Total T Cells: Change at Early Termination: number analyzed (Participants) | 1 | 0 | 1
  Total T Cells: Change at Early Termination | 350.0 |  | 393.0
  Total T Cells: Change at PT FU Week 24: number analyzed (Participants) | 1 | 0 | 0
  Total T Cells: Change at PT FU Week 24 | 220.0 |  |

9. Secondary Outcome: Change From Baseline in Urinary IgG, IgA, and IgM Levels
Description: Urinary IgG, IgA and IgM levels to be measured by Immuno-Electrophoresis.
Time Frame: Baseline (Day1), Weeks 24, 48 and Early Termination (up to earlier than Week 72)
Population: As per changed in planned analysis the outcome measure related to Urinary Immunoglobulins was not assessed.
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibody (ADA)
Description: Percentage of participants with positive ADA were reported.
Time Frame: Baseline up to safety follow-up (96 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
percentage of participants | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Clinical Significant Abnormalities in Laboratory Assessments
Description: Laboratory investigation included hematology, biochemistry, urinalysis and Urine sediment analysis. Clinical significance was to be decided by the investigator.
Time Frame: Baseline up to safety follow-up (96 weeks)
Population: As per changed in planned analysis the outcome measure related to clinically significant abnormalities in laboratory assessments was not assessed.
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Clinical Significant Abnormalities in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure, pulse rate, weight and height. The systolic and diastolic blood pressure and pulse rate was measured after the participants have in a rested at least 3 minutes in seated position. Clinical significance was to be decided by the investigator.
Time Frame: Baseline up to safety follow-up (96 weeks)
Population: As per changed in planned analysis the outcome measure related to clinically significant abnormalities in vital signs was not assessed.
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Clinical Significant Abnormalities in 12-Lead Electrocardiograms (ECGs)
Description: 12-lead ECG were recorded after the participants have rested for at least 15 minutes in supine position. Clinically significance was decided by the investigator. The number of participants with clinically significant abnormalities in 12-lead ECG were reported.
Time Frame: Baseline up to safety follow-up (96 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
Number analyzed (Participants) | 5 | 6 | 5
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to safety follow up period (96 weeks)
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 3/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Atacicept 25 mg (N=6) | Atacicept 75 mg (N=5)
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Atacicept 25 mg (N=6) | Atacicept 75 mg (N=5)
Injection site erythema (General disorders) | 0 | 4 | 1
Injection site bruising (General disorders) | 0 | 3 | 0
Injection site pruritus (General disorders) | 0 | 3 | 0
Injection site reaction (General disorders) | 0 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 1 | 0
Injection site inflammation (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to poor enrollment and Part B was not conducted as per Sponsor decision. This decision was not related to any safety or efficacy findings regarding Atacicept.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02808429/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT02808429/SAP_001.pdf